CLINICAL TRIAL: NCT06735911
Title: Assessment at 4.5 Months of the Effect of a Dermatology-Oriented Spa Therapy on the Quality of Life of Patients With Psoriasis (BAREGES)
Brief Title: Assessment of the Effect of a Dermatology-Oriented Spa Therapy on the Quality of Life of Patients With Psoriasis
Acronym: BAREGES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thermes de Bareges (Other)
Collaborators: Floralis (Industry); University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00700-47
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: psoriasis; spa therapy
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: before / after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: patient treated with a dermatology-oriented spa therapy (Experimental): Thermal treatments among the following: Filiform shower, simple bath, aerated bath, general shower, compresses, nebulization inhalation, multiple local mud applications, and drinking cure.
  Interventions: Other: Spa therapy

INTERVENTIONS:
Other: Spa therapy — Thermal treatments among the following: Filiform shower, simple bath, aerated bath, general shower, compresses, nebulization inhalation, multiple local mud applications, and drinking cure.
  Other Names: spa treatment; spa care

SUMMARY:
Evaluation of the effect of a dermatology-oriented spa therapy at 4.5 months on the quality of life of patients suffering from psoriasis

DETAILED DESCRIPTION:
BAREGES is a:

prospective, before/after, cohort follow-up study with repeated measurements monocentric study with the dispensation of a 3-week dermatolgy-oriented spa therapy in Barèges

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years Patient with psoriasis Stable treatment in the last 6 months. DLQI > 10 Patient presenting an indication for thermal treatment focused on dermatology (possible dual orientation).

Patient affiliated to the social security system or such a system Available for an 18-day spa treatment and a 9-month follow-up For women of childbearing age: effective contraception Patient information and informed consent signature

Exclusion Criteria:

Contraindication to thermal treatment (e.g., ongoing chemotherapy/radiotherapy, uncontrolled progressive neoplasia, progressive heart disease, etc., according to the investigator's assessment) Predictable intolerance to thermal treatments (intolerance to heat, baths, etc.) Patient who has already undergone a dermatology-oriented spa treatment within the current thermal season Subject already included in an interventional clinical research protocol Persons referred to in articles L1121-5 to L1121-8 of the "Code de la Santé Publique" (pregnant women, women in labour and parturient and nursing mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure or not being able to verbally communicate their agreement, minor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of a complete thermal treatment (moderate impact) for a dermatological indication on the quality of life of patients with psoriasis | 4.5 months
  Percentage of patients with a score ≤ 10 (moderate impact) on the Dermatology Life Quality Index (DLQI) questionnaire at 4.5 months.The DLQI score is between 0 and 30 where a high score indicates a significant impairment of quality of life.

SECONDARY OUTCOMES:
To evaluate the effect of a complete thermal treatment (low impact) for a dermatological indication on the quality of life of patients with psoriasis at 4.5 months, taking into account all the care provided | 4.5 months
  Percentage of patients with a score ≤ 5 (low impact) on the Dermatology Life Quality Index (DLQI) questionnaire at 4.5 months. The DLQI score is between 0 and 30 where a high score indicates a significant impairment of quality of life.
To evaluate dermatology-specific quality of life (quantitative DLQI score) | 4.5 and 9 months
  Comparison of the mean scores of the dermatology-specific quality of life questionnaire (DLQI) at inclusion (pre-thermal treatment), at 4.5 months (post-thermal treatment), and at 9 months after inclusion.The DLQI score is between 0 and 30 where a high score indicates a significant impairment of quality of life.
To evaluate overall quality of life using the EQ-5D-5L questionnaire. | 4.5 and 9 months
  Change in overall quality of life (EQ-5D-5L questionnaire) between inclusion, 4.5 months, and 9 months after inclusion.
  The EQ5D-5L essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  There are five dimensions assessed in the descriptive system: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. A higher score means better outcome.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. Score from 0 to 100. A higher score means better outcome.
To evaluate the clinical improvement of psoriasis in the short and medium term. | 4.5 and 9 months
  The PASI (Psoriasis Area and Severity Index) is a scale used to assess the clinical severity of psoriasis. The PASI will be measured at inclusion, 4.5 months, and 9 months.
  The minimum PASI score is 0, indicating no lesions. The maximum PASI score is 72, representing maximum involvement of all body areas with the highest severity.
To evaluate pain and pruritus. | 4.5 and 9 months
  A self-questionnaire (Visual Analog Scale) will be presented to the patients to measure pain and pruritus associated with skin lesions at inclusion, 4.5 months, and 9 months.
  These two results will be analyzed quantitatively. The minimum score is 0, indicating no pain or pruritus, while the maximum score is 10, representing the worst imaginable pain or intolerable pruritus.
Physician/Patient perception : The physician's and patient's opinion will be requested to assess the perceived benefit of the treatment. | 4.5 and 9 months
  This evaluation will be conducted at the investigator's office 4.5 months and 9 months after inclusion using a 5-point Likert scale.
Medication consumption | 4.5 and 9 months
  Collection of medication consumption to evaluate the benefit of the spa therapy (comparison of consumption before and after treatment)
Evolution of the general clinical criteria : Body Mass Index (BMI) | 4.5 and 9 months
  Comparison of the Body Mass Index between enrolment, and 4.5 months and 9 months after enrolment
Evolution of the general clinical criteria : systolic blood pressure | 4.5 and 9 months
  Comparison of the systolic blood pressure between enrolment, and 4.5 months and 9 months after enrolment
Evolution of the general clinical criteria : diastolic blood pressure | 4.5 and 9 months
  Comparison of the diastolic blood pressure between enrolment, and 4.5 months and 9 months after enrolment
Evolution of the general clinical criteria : heart rate | 4.5 and 9 months
  Comparison of the heart rate between enrolment, and 4.5 months and 9 months after enrolment
Evaluation of the use of care related or not to psoriasis at 4.5 and 9 months | 4.5 and 9 months
  Collection of medical events related or not to psoriasis (number of SAE, number of hospitalizations, number of medical and paramedical procedures)
Evaluation of compliance with the spa therapy | 3 weeks
  Comparison of the thermal treatments received by the patient during the spa therapy with the thermal treatments prescribed by the thermal doctor at the start of the spa therapy, collected in the spa treatment booklet

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Cabinet Luz Saint Sauveur, Pierrefitte-Nestalas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebwohl M, Ellis C, Gottlieb A, Koo J, Krueger G, Linden K, Shupack J, Weinstein G. Cyclosporine consensus conference: with emphasis on the treatment of psoriasis. J Am Acad Dermatol. 1998 Sep;39(3):464-75. doi: 10.1016/s0190-9622(98)70325-1. PMID 9738783
- [Background] SOLOMON WM, NETHERTON EW, NELSON PA, ZEITER WJ. Treatment of psoriasis with Goeckerman technic. Arch Phys Med Rehabil. 1955 Feb;36(2):74-7. No abstract available. PMID 13229486
- [Background] Kazandjieva J, Grozdev I, Darlenski R, Tsankov N. Climatotherapy of psoriasis. Clin Dermatol. 2008 Sep-Oct;26(5):477-85. doi: 10.1016/j.clindermatol.2008.05.001. PMID 18755366